CLINICAL TRIAL: NCT00579462
Title: Methylated Genes in Blood as Biomarkers for Advanced Lung Cancer
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); University of Southern California (Other)
Responsible Party: Christopher Azzoli, Memorial Sloan-Kettering Cancer Center
Other Study IDs: 02-111
Record Dates: First submitted 2007-12-19; First posted 2007-12-24 (Estimated); Last update posted 2010-12-01 (Estimated); Status verified 2010-11

CONDITIONS: Lung Cancer
Keywords: Stage III or IV Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients with advanced lung cancer.
  Interventions: Other: Blood and Tissue studies

INTERVENTIONS:
Other: Blood and Tissue studies — Blood will be collected from participating patients at baseline, as close as possible to the date of their baseline radiologic assessment. Three follow-up blood collections will be drawn, each within 7-10 days of each follow-up radiologic evaluation.

SUMMARY:
The purpose of this study is to study whether the presence of lung cancer in your body can be detected by testing the blood, and if the results of these blood tests change as your tumor shrinks or grows.

DETAILED DESCRIPTION:
This is a cooperative research project involving patients on the Thoracic Oncology Service at Memorial Sloan-Kettering Cancer Center, and the laboratory of Dr. Peter Danenberg, Professor of Biochemistry and Molecular Biology, University of Southern California / Norris Comprehensive Cancer Center in Los Angeles, California. The primary objectives are to measure the proportion of patients with advanced (stage III-IV) lung cancer with methylated genes in their blood, and to determine if response to chemotherapy (complete or partial radiologic response) in patients with advanced lung cancer renders methylated genes undetectable in the blood. This research project will enroll approximately 80 patients per year over 4 years to generate a sample size of approximately 320 patients.Blood will be collected from participating patients at baseline, as close as possible to the date of their baseline radiologic assessment. Three follow-up blood collections will be drawn, each within 7-10 days of each follow-up radiologic evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven advanced (stage III-IV) lung cancer
* Measurable and/or evaluable disease
* Enrollment in an MSKCC protocol of experimental chemotherapy with radiologic response rate as an efficacy outcome variable, or prescription of standard chemotherapy in which the patient will be receiving routine radiological scans (every 4-8 weeks) as standard clinical practice.
* Signed written informed consent

Exclusion Criteria:

-None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients being seen in Thoracic Oncology Clinic
Sampling Method: Non-Probability Sample
Enrollment: 281 (Actual)
Dates: Start 2003-01; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
To measure the proportion of patients with advanced (stage IIIB/IV) lung cancer with methylated genes in their blood and determine if response to chemotherapy (CR or PR radiologic response) renders methylated genes undetectable in blood. | 1 year

SECONDARY OUTCOMES:
To collect data regarding time to disease progression in order to explore whether pretreatment and/or posttreatment blood levels of methylated genes are associated with an increased chance of disease progression. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Azzoli, M.D., Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Related Info — http://www.mskccc.org